CLINICAL TRIAL: NCT02473705
Title: Pathways to Improving Functional Capacity in Older Patients With Chronic Kidney Disease and Cardiovascular Disease
Acronym: CKD&CAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find eligible participants to participate in the study.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WakeForest
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2016-09

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease
Keywords: Geriatric; bicarbonate; omega polyunsaturated fatty acids; exercise capacity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases | interventions — Fish Oils; Bicarbonates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fish Oil and Bicarbonate placebo (Active Comparator): 1280mg of fish oil per day and bicarbonate placebo
  Interventions: Dietary Supplement: Fish Oil and Bicarbonate Placebo
- Fish Oil Placebo and Bicarbonate (Active Comparator): fish oil placebo and 1mg of bicarbonate per Kg of body weight per day
  Interventions: Dietary Supplement: Fish Oil Placebo and Bicarbonate
- Fish Oil and Bicarbonate (Experimental): 1280mg of fish oil per day and 1mg of bicarbonate per Kg of body weight per day
  Interventions: Dietary Supplement: Fish Oil and Bicarbonate
- Fish Oil placebo and Bicarbonate placebo (Placebo Comparator): Fish oil placebo and Bicarbonate placebo
  Interventions: Dietary Supplement: Fish Oil Placebo and Bicarbonate Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil and Bicarbonate — 1280mg of fish oil per day and 1mg of bicarbonate per Kg of body weight per day
  Other Names: Nordic Naturals - Ultimate Omega
  Arms: Fish Oil and Bicarbonate
Dietary Supplement: Fish Oil and Bicarbonate Placebo — 1280mg of fish oil per day and bicarbonate placebo (Methylcellulose)
  Other Names: Nordic Naturals - Ultimate Omega
  Arms: Fish Oil and Bicarbonate placebo
Dietary Supplement: Fish Oil Placebo and Bicarbonate — Fish oil placebo (soybean oil) and 1mg of bicarbonate per Kg of body weight per day
  Arms: Fish Oil Placebo and Bicarbonate
Dietary Supplement: Fish Oil Placebo and Bicarbonate Placebo — Fish oil placebo (soybean oil) and bicarbonate placebo (Methylcellulose)
  Arms: Fish Oil placebo and Bicarbonate placebo

SUMMARY:
The purpose of this research study is to study the effect of fish oil and bicarbonate (baking soda) on exercise. In this study fish oil, bicarbonate or both will be compared to placebo to see if study participants increase exercise capacity.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) have a high morbidity and mortality from cardiovascular disease (CVD). Both conditions are common in older patients. Reduced exercise capacity predicts poorer outcomes in patients with CVD2 and CKD. Although exercise tolerance is impaired in CKD4 limited improvement in these patients is possible. A critical gap in knowledge is how to optimize exercise capacity in these patients to improve quality and possibly length of life.

In CKD, both structure and function of skeletal muscle are deranged. In addition, energy production by mitochondria which falls with age, and various diseases is also reduced in CKD. Recent studies from our group have reported that differences in mitochondrial function are associated with variances in physical ability, exercise capacity, and gait speed.

In preliminary data, patients entering our Cardiac Rehabilitation (CR) with Stage III CKD [glomerular filtration rate (GFR) of <60 ml/min/1.73 m2] had a decreased improvement in exercise capacity compared to those with a normal GFR (Δ1.7 vs 2.7 Metabolic Equivalents of Exercise or METs, p<0.05) despite the same degree of adherence. Exercise capacity after CR in patients with a reduced GFR was greater in n-3 polyunsaturated fatty acids (n-3 PUFA) users than in non-users [Δ MET 2.0 (1.4-2.5) vs 1.4 (1.1-1.7), p<0.05], suggesting that n-3 PUFA with exercise may be better than exercise alone. With beneficial clinical effects in CKD, n-3 PUFA are now being extensively investigated in the dialysis population. In other patient populations, including those with chronic obstructive pulmonary disease and dilated cardiomyopathy daily ingestion/use of n-3 polyunsaturated fatty acids (n-3 PUFA) or fish oil improves exercise capacity. This intervention is safe, simple and well-tolerated. Multiple lines of evidence suggest muscle and mitochondrial function improve with exercise and n-3 PUFA supplementation.Such treatment may improve mitochondrial bioenergetics by various mechanisms including up-regulation of mitochondrial biogenesis and genes involved in mitochondrial fatty acid oxidation, as well as increase in mitochondrial content, and function. Flow mediated vasodilation is impaired in CKD. It too may be improved by n-3 PUFA supplementation which could be an alternative mechanism for improved oxygen delivery to muscle in older patients with CAD and CKD as in the non-CKD population. A further possible benefit of n-3 PUFA is suppression of inflammation.

Current practice, however, is to enter patients with CAD and CKD into standard CR without prescription of n-3 PUFA.

Experimental and epidemiological studies indicate that acidemia and metabolic acidosis are associated with the development and progression of CKD and with increased mortality in these patients. Metabolic acidosis associated with CKD also contributes to skeletal muscle atrophy by activation of the ubiquitin-proteasome axis. Even slight correction of acidosis can improve the anabolic state of muscle by downregulation of the ubiquitin-proteasome system. Clinically, bicarbonate supplementation may improve muscle function. This intervention is also safe, simple and well-tolerated.

Given that muscular function is abnormal in CKD and that both n-3 PUFA and bicarbonate supplementation have been shown to improve muscular function and exercise capacity, it is our purpose in this investigation to study the effects of these substances on exercise capacity in patients with CAD and CKD.

The investigators propose a double-blind, placebo-controlled, randomized, 2x2 factorial design, pilot study of n-3 PUFA and/or oral bicarbonate use in older (age >60 years) CAD patients with concomitant CKD enrolling in a standard, 3-month CR program. The investigators will assess the effects of this intervention on exercise capacity, markers of inflammation and serum bicarbonate concentration. The investigator's goal is to obtain 8 evaluable patients per group. Exercise capacity will be measured by Oxygen (VO2) peak. Response to bicarbonate will be monitored by serum bicarbonate concentration. Since CKD may adversely affect muscle function both by acidosis and/or mitochondrial function, the investigator's propose that these may be mechanisms for the poorer exercise capacity in these patients. The investigator's overarching hypothesis is that exercise capacity response to CR in older patients with CKD may be modifiable by concomitant n-3 PUFA and/or bicarbonate use to suppress acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Referred to Cardiac Rehabilitation after acute coronary syndromes or percutaneous intervention
* Stage III Chronic kidney disease
* Clinically stable with no mobility conditions that preclude safe walking and able to walk
* No contraindications that will prevent measurement of physical ability and exercise capacity including severe arthritis or musculoskeletal disorders
* knee/hip replacement or spinal surgery in past year
* Approved for participation by Principal Investigator
* Not involved in any other research study or undergoing physical therapy
* Able to provide own transportation to study visits and intervention
* Willing to provide written consent

Exclusion Criteria:

* Currently taking fish oil supplements
* Advanced malignancy or other medical condition with life expectancy less than 2 years or undergoing active chemotherapy or radiation therapy
* Oxygen-dependent chronic obstructive pulmonary disease
* Normal kidney function or advanced chronic kidney disease (glomerular filtration rate < 20 mL/min/1.73 m2, on dialysis or dialysis anticipated within 6 months)
* Mini-mental state examination score of ≤ 21 or previously diagnosed dementia or cognitive impairment limiting ability to participate in rehabilitation and follow study protocols
* Chronic anemia with hemoglobin <10 gm/dl for males, <9 gm/dl for females or acute anemia requiring transfusion
* Significant impairment from a prior stroke or other neurologic disease or injury that would preclude participation
* Severe peripheral arterial disease that is the primary limitation to ambulation
* Medical condition that would limit exercise
* High risk for non-adherence as determined by screening evaluation
* Patients who have undergone renal transplantation
* Currently taking bicarbonate supplementation
* Current or recent (within the last 3 months) participation in an exercise program
* Carbon Dioxide level greater than the middle of the normal range i.e. 27mmol/L and thus predisposing to metabolic alkalosis
* Moderate 2+ or greater lower extremity edema
* Active congestive heart failure
* Ejection fraction less than 35%
* Patients using walkers and canes

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of VO2 peak at 12 weeks | 12 weeks
  Treadmill during a graded exercise test to exhaustion using a Ramp protocol

CONTACTS AND LOCATIONS:
Overall Officials: Killian Robinson, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health Cardiac Rehab, Winston-Salem, North Carolina, United States